CLINICAL TRIAL: NCT03182153
Title: Extended Ambulatory Monitoring Improves Risk Stratification in Hypertrophic Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Other Study IDs: SEEQ
Record Dates: First submitted 2017-05-30; First posted 2017-06-09 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Enrolled subjects: Subjects who are diagnosed with HCM and require routine extended cardiac monitoring for risk stratification of sudden cardiac death. All subjects will receive 28 days of external cardiac monitoring.
  Interventions: Device: Extended Cardiac Monitoring

INTERVENTIONS:
Device: Extended Cardiac Monitoring — Extended External Cardiac Monitoring
  Other Names: Medtronic SEEQ™ Mobile Cardiac Telemetry

SUMMARY:
Eligible subjects will wear 4 consecutive external monitoring devices for a total of 28 days of monitoring.

DETAILED DESCRIPTION:
Eligible subjects will be monitored with a SEEQ device. The SEEQ device is a patch-like device that is worn externally on the chest and continuously monitors heart rhythm. Each device is worn for seven days and replaced with additional devices for a total of 28 days of monitoring. Subjects will return the SEEQ equipment at the end of the monitoring period. Subjects will be contacted by telephone or seen at the clinic approximately 60 days from the first day of monitoring. Information will be gathered about medications and any cardiac interventions the subject may have had.

Subjects will again be contacted by telephone or seen in the clinic approximately 1 year from study start. Information will be gathered about general health, changes in medications, and cardiac interventions or events. Cardiac testing results will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of HCM Scheduled for routine ambulatory monitoring for risk stratification Followed at the Chanin T. Mast HCM Center at Morristown Medical Center

Exclusion Criteria:

Prior implantation of an ICD History of persistent/permanent atrial fibrillation (AF)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any HCM patient followed in the Chanin T. Mast HCM Center at Morristown Medical Center, Morristown, NJ, who is prescribed holter monitoring for risk stratification for SD.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12-28 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk Stratification for sudden death (SD) | Through study completion, an average of 1 year.
  We aim to determine if longer term monitoring (28 days) with the Medtronic SEEQ MCT device identifies a greater burden of non-sustained ventricular tachycardia (NSVT) compared to conventional shorter monitoring periods (48 hours), and thereby potentially identify a subset of HCM patients who may be at higher risk of SD and benefit from a primary prevention implantable cardioverter-defibrillator (ICD) .

SECONDARY OUTCOMES:
Detection of Atrial Fibrillation | Through study completion, an average of 1 year.
  To determine if longer term monitoring (28 days) with the Medtronic SEEQ MCT device identifies a greater burden of symptomatic (or asymptomatic) atrial fibrillation compared to conventional shorter monitoring periods (48 hours), and thereby identify a subset of HCM patients who may be at higher risk of symptom progression and stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No